CLINICAL TRIAL: NCT05228340
Title: The Efficacy of Flexor Tenotomy on the Prevention of Recurrent Diabetic Foot Ulcers: a Randomized Controlled Trial
Brief Title: Flexor Tenotomy and Ulcer Recurrence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Marieke Mens, Coördinating investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL78504.018.21
Record Dates: First submitted 2022-01-11; First posted 2022-02-08 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Hammer Toe Syndrome; Foot Ulcer, Diabetic
MeSH Terms: conditions — Hammer Toe Syndrome; Diabetic Foot

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Flexor tenotomy
  Interventions: Procedure: Flexor tenotomy
- Controle (No Intervention): Usual-care

INTERVENTIONS:
Procedure: Flexor tenotomy — Minimally-invasive percutaneous needle flexor tenotomy of the long digital flexor tendon
  Arms: Intervention

SUMMARY:
The main purpose of this study is to assess the efficacy of flexor tenotomy on the prevention of recurrence of toe ulcers in people with diabetes and a history of toe ulceration. Additionally, the investigators aim to assess interphalangeal joints (IPJ) and metatarsophalangeal joint (MTPJ) angles in a weight-bearing and non-weight-bearing position, bare-foot plantar pressure during walking and quality of life before and after the intervention and compare between study groups.

DETAILED DESCRIPTION:
Foot ulcers are a frequent problem in patients with diabetes mellitus and can lead to amputations. Prevention of these ulcers is therefore of paramount importance. Claw/hammer toe deformity is commonly seen in patients with diabetes. These deformities increase the risk of ulcer development specifically at the (apex of) the toe. Tenotomy of the tendon of the flexor muscles of the toes (tendon tenotomy) can be used to treat the consequences of claw/hammer toe deformity with the goal to prevent ulcer recurrence. For indication and assessment of outcomes of flexor tenotomy, weight-bearing CT and dynamic barefoot plantar pressure measurement can be used. This mono-center investigator blinded randomized controlled trial will compare the flexor tenotomy with usual care (including orthoses and shoe offloading). The effect on ulcer recurrence, toe joint angles, barefoot plantar pressure and quality of life will be assessed and compared between the intervention and control group.

ELIGIBILITY:
Inclusion Criteria:

* A minimum age of 18 years
* Sufficient understanding of Dutch/English language
* Capable of filling out informed consent
* Peripheral polyneuropathy
* Diabetes mellitus type 1 or 2
* A minimum of one claw/hammer toe
* A documented history of diabetic ulcers underneath the toe apex in the past 5 years

Exclusion Criteria:

* No written informed consent
* Not meeting the inclusion criteria
* Open ulcers on the toes
* Previous participation in the study
* Pregnant women
* Concomitant participation in a study in which the patient is exposed to X-rays

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Ulcer recurrence | 24 months
  Ulcer recurrence on the toe, adjacent toe, and metatarsal heads

SECONDARY OUTCOMES:
DIPJ, PIPJ and MTPJ angles | Baseline, 6 and 12 months
  DIPJ, PIPJ and MTPJ angles during weight-bearing and non-weight-bearing
Barefoot pressure pattern | Baseline, 6 and 12 months
  Barefoot pressure pattern
Patient-reported outcome measures: EuroQol's EQ-5D-5L | Baseline, 6, 12 and 24 months
  Quality of life determined by EQ-5D-5L
Patient-reported outcome measures: SF-36 | Baseline, 6, 12 and 24 months
  Quality of life determined by SF-36
Incremental cost-effectiveness in QALY's of flexor tenotomy after 2 years | 24 months
  Cost-effectiveness of additional flexor tenotomy compared to usual-care only

CONTACTS AND LOCATIONS:
Overall Officials: Gino M.M.J. Kerkhoffs, MD, PhD, Principal Investigator — Amsterdam University Medical Centers
Locations (1):
- Amsterdam UMC - location MAMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mens MA, Busch-Westbroek TE, Bus SA, van Netten JJ, Wellenberg RHH, Streekstra GJ, Maas M, Nieuwdorp M, Kerkhoffs GMMJ, Stufkens SAS. The efficacy of flexor tenotomy to prevent recurrent diabetic foot ulcers (DIAFLEX trial): Study protocol for a randomized controlled trial. Contemp Clin Trials Commun. 2023 Mar 11;33:101107. doi: 10.1016/j.conctc.2023.101107. eCollection 2023 Jun. PMID 36950303